CLINICAL TRIAL: NCT02888054
Title: A Phase 1, Randomized, Open-Label, Replicate, Crossover Study to Assess the Bioequivalence of Lesinurad/Allopurinol Fixed-Dose Combination Tablets and Coadministered Lesinurad and Allopurinol Tablets in Fed Healthy Adult Subjects
Brief Title: Lesinurad/Allopurinol 200/300 FDC Tablets Bioequivalence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RDEA594-503
Record Dates: First submitted 2016-08-30; First posted 2016-09-02 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Healthy
MeSH Terms: interventions — lesinurad; Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence ABBA (Experimental): Day 1: lesinurad/allopurinol 200/300 FDC tablet (Sequence A) Day 8: coadministered lesinurad 200 mg + allopurinol 300 mg tablets (Sequence B) Day 15: coadministered lesinurad 200 mg + allopurinol 300 mg tablets (Sequence B) Day 22: lesinurad/allopurinol 200/300 FDC tablet (Sequence A)
  Interventions: Drug: lesinurad/allopurinol 200/300 FDC tablet; Drug: lesinurad 200 mg; Drug: allopurinol 300 mg
- Sequence BABA (Experimental): Day 1: coadministered lesinurad 200 mg + allopurinol 300 mg tablets (Sequence B) Day 8: lesinurad/allopurinol 200/300 FDC tablet (Sequence A) Day 15: coadministered lesinurad 200 mg + allopurinol 300 mg tablets (Sequence B) Day 22: lesinurad/allopurinol 200/300 FDC tablet (Sequence A)
  Interventions: Drug: lesinurad/allopurinol 200/300 FDC tablet; Drug: lesinurad 200 mg; Drug: allopurinol 300 mg
- Sequence ABAB (Experimental): Day 1: lesinurad/allopurinol 200/300 FDC tablet (Sequence A) Day 8: coadministered lesinurad 200 mg + allopurinol 300 mg tablets (Sequence B) Day 15: lesinurad/allopurinol 200/300 FDC tablet (Sequence A) Day 22: coadministered lesinurad 200 mg + allopurinol 300 mg tablets (Sequence B)
  Interventions: Drug: lesinurad/allopurinol 200/300 FDC tablet; Drug: lesinurad 200 mg; Drug: allopurinol 300 mg
- Sequence BAAB (Experimental): Day 1: coadministered lesinurad 200 mg + allopurinol 300 mg tablets (Sequence B) Day 8: lesinurad/allopurinol 200/300 FDC tablet (Sequence A) Day 15: lesinurad/allopurinol 200/300 FDC tablet (Sequence A) Day 22: coadministered lesinurad 200 mg + allopurinol 300 mg tablets (Sequence B)
  Interventions: Drug: lesinurad/allopurinol 200/300 FDC tablet; Drug: lesinurad 200 mg; Drug: allopurinol 300 mg

INTERVENTIONS:
Drug: lesinurad/allopurinol 200/300 FDC tablet
Drug: lesinurad 200 mg
Drug: allopurinol 300 mg

SUMMARY:
This study will assess the bioequivalence (BE) of Lesinurad/Allopurinol Fixed-Dose Combination (FDC) Tablets and Coadministered Lesinurad and Allopurinol Tablets in Fed Healthy Adult Subjects

DETAILED DESCRIPTION:
The study will assess the BE between lesinurad/allopurinol 200/300 FDC tablets and coadministered lesinurad and allopurinol tablets in the fed state.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index ranging between 18 kg/m2 and 30 kg/m2.
* Screening serum urate level is ≤ 7.0 mg/dL.

Exclusion Criteria:

* Asian subject who has a positive test for the HLA-B*5801 allele.
* History or suspicion of kidney stones.
* Estimated creatinine clearance, as determined at Screening, of < 90 mL/min calculated by the Cockcroft-Gault formula using ideal body weight.
* Undergone major surgery within 3 months prior to Screening.
* Donated blood or experienced significant blood loss (> 450 mL) within 12 weeks prior to Day 1or has given a plasma donation within 4 weeks prior to Day 1.
* Inadequate venous access or unsuitable veins for repeated venipuncture.
* Received any strong or moderate enzyme-inducing drug or product within 2 months prior to Screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2016-10-18 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) endpoints in terms of maximum observed concentration (Cmax) for lesinurad/allopurinol 200/300 FDC tablets relative to lesinurad and allopurinol coadministered monocomponent tablets | Days 1, 8, 15, and 22
  Cmax is the maximum observed concentration of a drug after administration
PK endpoints in terms of time of occurrence of maximum observed concentration (tmax) for lesinurad/allopurinol 200/300 FDC tablets relative to lesinurad and allopurinol coadministered monocomponent tablets | Days 1, 8, 15, and 22
  Tmax is the time of occurrence of cmax
PK endpoints in terms of area under plasma concentration time curve from zero to the last quantifiable sampling timepoint (AUC last) for lesinurad/allopurinol 200/300 FDC tablets relative to lesinurad and allopurinol coadministered monocomponent tablets | Days 1, 8, 15, and 22
  AUC last is a measure of total plasma concentration from time zero to the last measurable concentration
PK endpoints in terms of area under the plasma concentration time curve from and from zero to infinity (AUC 0-∞) for lesinurad/allopurinol 200/300 FDC tablets relative to lesinurad and allopurinol coadministered monocomponent tablets | Days 1, 8, 15, and 22
  AUC 0-∞ is a measure of total concentration from time zero to infinity
PK endpoints in terms of apparent terminal half-life (t1/2) for lesinurad/allopurinol 200/300 FDC tablets relative to lesinurad and allopurinol coadministered monocomponent tablets | Days 1, 8, 15, 22
  t1/2 is a measure of apparent terminal half-life

SECONDARY OUTCOMES:
Incidence of Adverse Events in terms of changes in laboratory parameters | 8 weeks
Incidence of Adverse Events in terms of electrocardiogram parameters | 8 weeks
Incidence of Adverse Events in terms of vital signs | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: N. Bhakta, Study Director — Ardea Biosciences, Inc.
Locations (1):
- Austin, Texas, United States